CLINICAL TRIAL: NCT03329573
Title: Randomized, Open Label, 2-way Crossover, Single Dose Bioequivalence Study of Paroxetine IR Tablets Manufactured in GSKT and Mississauga Sites in Healthy Chinese Participants Under Fasting and Fed Conditions
Brief Title: Bioequivalence Study of Paroxetine Immediate Release (IR) Tablets Manufactured in GlaxoSmithKline Tianjin (GSKT) and Mississauga Sites in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 207652
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Results first posted 2019-08-19 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Anxiety Disorders
Keywords: Cross-over; Chinese; GSKT; Mississauga; Healthy; Bioequivalence; Paroxetine
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: In this study, each subject will receive paroxetine IR 40mg A or B in a cross-over manner
Masking Description: This study is an open-label treatment period; hence, masking will not be performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- AB treatment sequence receivers in fasting group (Experimental): Eligible subjects will receive a single dose of Paroxetine IR tablets A in Period 1 followed by Paroxetine IR tablets B in Period 2 in fasting state.
  Interventions: Drug: Paroxetine IR tablets A; Drug: Paroxetine IR tablets B
- BA treatment sequence receivers in fasting group (Experimental): Eligible subjects will receive a single dose of Paroxetine IR tablets B in Period 1 followed by Paroxetine IR tablets A in Period 2 in fasting state.
  Interventions: Drug: Paroxetine IR tablets A; Drug: Paroxetine IR tablets B
- AB treatment sequence receivers in fed group (Experimental): Eligible subjects will receive a single dose of Paroxetine IR tablets A in Period 1 followed by Paroxetine IR tablets B in Period 2 in fed state.
  Interventions: Drug: Paroxetine IR tablets A; Drug: Paroxetine IR tablets B
- BA treatment sequence receivers in fed group (Experimental): Eligible subjects will receive a single dose of Paroxetine IR tablets B in Period 1 followed by Paroxetine IR tablets A in Period 2 in fed state.
  Interventions: Drug: Paroxetine IR tablets A; Drug: Paroxetine IR tablets B

INTERVENTIONS:
Drug: Paroxetine IR tablets A — Paroxetine IR tablets A will be the investigational drug. These are film coated tablets with unit dose strength of 20 milligrams (mg) and will be administered via oral route. These tablets will be manufactured in GSKT.
Drug: Paroxetine IR tablets B — Paroxetine IR tablets B will be the reference drug. These are film coated tablets with unit dose strength of 20 mg and will be administered via oral route. These tablets will be manufactured in Mississauga.

SUMMARY:
Paroxetine is a selective serotonin reuptake inhibitor (SSRI) and paroxetine IR tablets have been approved for the treatment of three anxiety indications in China. This bioequivalence study will evaluate Paroxetine IR tablets manufactured in GSKT (A) and Mississauga (B) sites in healthy Chinese subjects under fasting and fed conditions to support the quality consistency evaluation. This is a single dose, open-label, randomized, two-period crossover study and will include a screening period (up to 7 days), two open-label treatment periods (up to 16 days) and a follow-up phase (up to 14 days after last-dose). The whole study will be divided into two groups, one for fasting condition enrolling approximately 36 subjects and another for fed condition for which approximately 44 subjects will be enrolled. In both groups, eligible subjects will be randomized to receive single dose of Paroxetine IR tablets A or B in a cross-over manner.

ELIGIBILITY:
Inclusion Criteria:

* Able to actively communicate with the investigator and to complete the study-related documents; able to understand the contents of the Informed consent form (ICF) and to sign a written ICF prior to any study-specific procedures.
* Males and females aged between 18 and 45 years inclusive, at the time of signing the informed consent.
* Non-smoking healthy males and females as assessed by medical history and physical examination. Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring. A subject with a clinical abnormality or laboratory parameters which are not specifically listed in the inclusion or exclusion criteria, outside the reference range for the population being studied may be included only if the Investigator (in consultation with the GSK Medical Monitor if necessary) agree and document that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures.
* Body weight>=50 kilograms (kg) (male) or 45kg(female) and Body mass index (BMI) 19.0 to 26.0 kg per meter square (kg/m^2) (inclusive).
* A female subject is eligible to participate if she is of: Child-bearing potential with negative pregnancy test as determined by serum or urine human chorionic gonadotropin (hCG) test at screening or prior to dosing and agrees to use the one of the defined contraception method during the study and until follow up contact.
* Male Subjects with female partners of child-bearing potential must agree to use one of the defined contraception methods during the study and until follow up contact.
* ALT, ALP and total bilirubin <=1.5x upper limit of normal (ULN) (isolated bilirubin >1.5x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent).
* Based on single or averaged corrected QT interval (QTc) values of triplicate ECGs obtained over a brief recording period: QTc < 450 milliseconds (msec); or QTc < 480 msec in subjects with bundlebranch block.

Exclusion Criteria:

* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Drug or alcohol abuse or dependency within one year prior to enrolment. History of regular alcohol consumption within one year of the study defined as: an average weekly intake of >14 drinks. One drink is equivalent to 12 grams (g) of alcohol: 12 ounces [360 milliliter (mL)] of beer, 5 ounces (150 mL) of wine or 1.5 ounces (45 mL) of 80 proof distilled spirits.
* Unstable disease conditions; any laboratory measurements assessed by the investigator as clinically relevant (including ECG, hematology, biochemistry and urine analysis, etc.)；any disorder that might interfere with the absorption, distribution, metabolism or excretion of the study drug; or in the investigator's opinion the disease may lead to safety concerns or interfere with the pharmacokinetics assessment.
* Subjects with concurrent or previous neuropsychological disorders, as assessed by Columbia Suicide Severity Rating Scale or by the investigator, have suicidal tendency, or have committed suicidal behavior/attempt.
* Known history of cerebral trauma, previous cerebral disorders, seizures or eating disorder, and other conditions that in the investigator's opinion may increase the risk of seizures.
* Exposure to more than four new chemical entities within 12 months prior to the first dosing day.
* Unable to refrain from the use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study medication.
* In subjects with concomitant use of monoamine oxidase inhibitors (MAOIs) (including linezolid, an antibiotic which is a reversible non-selective MAOIs and methylthioninium chloride (methylene blue)) or within two weeks of terminating treatment with MAOIs.
* In subjects with concomitant use of thioridazine or pimozide.
* The subject has participated in a clinical trial and has received an investigational product within 90 days prior to the first dosing day in the current study, or has participated in a clinical trial without receiving any investigational product within 30 days prior to the first dosing day in the current study.
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months.
* Serum human immuno-deficiency virus (HIV) antibody or Syphilis antibody positive.
* A positive pre-study drug/alcohol screen.
* Known allergy to paroxetine IR Tablets or any of its components.
* Blood donation in excess of 400 mL in the 3 months prior to enrolment.
* Obvious evidence of active hematological diseases, or significant blood loss in the last 3 months. History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Lactating females or women of child bearing potential used oral or implanted contraceptives within the 30 days prior to enrolment, or received injections of chronically acting contraceptives in the 1 year prior to study initiation.
* Other conditions which, in the Investigator's judgment, render subjects unsuitable for the clinical study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-08-03 (Actual); Study Completion 2018-08-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=20306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a single dose, open-label, randomized, two-period crossover study to demonstrate the bioequivalence of Paroxetine immediate release (IR) tablets manufactured in GlaxoSmithKline Tianjin (GSKT) (A) and Mississauga (B) sites in healthy Chinese participants under fasting and fed conditions.
Pre-assignment Details: Participants received treatment in one of the two sequences; treatment A (GSKT, Paroxetine IR investigational drug) followed by treatment B (Mississauga, Paroxetine IR reference drug) or vice versa in each of the treatment period 1 and 2. A total of 85 (47 under fed condition and 38 under fasting condition) participants were enrolled.
Groups:
- Paroxetine 40 mg, GSKT Followed by Mississauga- Fed: Eligible participants received a single dose of treatment A: GSKT, Paroxetine IR 40 milligrams (mg) (20 mg*2 tablets) administered orally on Day 1 in treatment period 1. It was followed by a washout period from Day 6 to Day 11. Participants received treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 12 in treatment period 2. All these doses were administered under fed condition.
- Paroxetine 40 mg, Mississauga Followed by GSKT- Fed: Eligible participants received a single dose of treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in treatment period 1. It was followed by a washout period from Day 6 to Day 11. Participants received treatment A: GSKT, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 12 in treatment period 2. All these doses were administered under fed condition.
- Paroxetine 40 mg, GSKT Followed by Mississauga- Fasted: Eligible participants received a single dose of treatment A: GSKT, Paroxetine IR 40 milligrams (mg) (20 mg*2 tablets) administered orally on Day 1 in treatment period 1. It was followed by a washout period from Day 6 to Day 11. Participants received treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 12 in treatment period 2. All these doses were administered under fasting condition.
- Paroxetine 40 mg, Mississauga Followed by GSKT- Fasted: Eligible participants received a single dose of treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in treatment period 1. It was followed by a washout period from Day 6 to Day 11. Participants received treatment A: GSKT, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 12 in treatment period 2. All these doses were administered under fasting condition.
Period: Treatment Period 1 (Up to 5 Days)
Arm/Group | Paroxetine 40 mg, GSKT Followed by Mississauga- Fed | Paroxetine 40 mg, Mississauga Followed by GSKT- Fed | Paroxetine 40 mg, GSKT Followed by Mississauga- Fasted | Paroxetine 40 mg, Mississauga Followed by GSKT- Fasted
Started | 23 | 24 | 19 | 19
Completed | 22 | 21 | 19 | 19
Not Completed | 1 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Period: Washout Period (Day 6 to Day 11)
Arm/Group | Paroxetine 40 mg, GSKT Followed by Mississauga- Fed | Paroxetine 40 mg, Mississauga Followed by GSKT- Fed | Paroxetine 40 mg, GSKT Followed by Mississauga- Fasted | Paroxetine 40 mg, Mississauga Followed by GSKT- Fasted
Started | 22 | 21 | 19 | 19
Completed | 22 | 21 | 19 | 19
Not Completed | 0 | 0 | 0 | 0
Period: Treatment Period 2 (Day 12 to Day 26)
Arm/Group | Paroxetine 40 mg, GSKT Followed by Mississauga- Fed | Paroxetine 40 mg, Mississauga Followed by GSKT- Fed | Paroxetine 40 mg, GSKT Followed by Mississauga- Fasted | Paroxetine 40 mg, Mississauga Followed by GSKT- Fasted
Started | 22 | 21 | 19 | 19
Completed | 21 | 20 | 19 | 19
Not Completed | 1 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paroxetine 40 mg, GSKT Followed by Mississauga- Fed | Paroxetine 40 mg, Mississauga Followed by GSKT- Fed | Paroxetine 40 mg, GSKT Followed by Mississauga- Fasted | Paroxetine 40 mg, Mississauga Followed by GSKT- Fasted | Total
Number analyzed (Participants) | 23 | 24 | 19 | 19 | 85
Age, Continuous [Mean (Standard Deviation); unit: Years] | 30.3 (7.53) | 27.1 (5.63) | 25.4 (5.86) | 28.1 (6.17) | 27.3 (6.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 10 | 9 | 10 | 40
  Male | 12 | 14 | 10 | 9 | 45
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian - East Asian Heritage | 23 | 24 | 19 | 19 | 85

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero Extrapolated to Infinite Time (AUC[0-infinity]) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated time points. Pharmacokinetic (PK) parameters of Paroxetine were calculated using non-compartmental methods. Statistical analysis of PK parameters was done using mixed effect model for evaluation of bioequivalence (BE). Point estimate and associated adjusted 90% confidence interval (CI) of difference between both the treatments were provided for AUC(0-infinity).
Time Frame: Pre-dose, 0.5 hour, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 7 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours, 72 hours and 96 hours post-dose in each treatment period
Population: BE analysis Population. BE analysis Population comprised of all randomized participants who completed all the planned treatments and provided at least one evaluable primary PK parameter data from both period 1 and period 2. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (90% Confidence Interval); unit: Hour*nanogram per milliliter
Groups:
- Paroxetine 40 mg, GSKT- Fed: Eligible participants received a single dose of treatment A: GSKT, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in either treatment period 1 or 2 as per randomization under fed condition.
- Paroxetine 40 mg, Mississauga- Fed: Eligible participants received a single dose of treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in either treatment period 1 or 2 as per randomization under fed condition.
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 40 | 40
Hour*nanogram per milliliter | 860.54 [728.07 to 1017.12] | 812.49 [687.42 to 960.33]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fed vs Paroxetine 40 mg, Mississauga- Fed; Test type: Equivalence — The two formulations were considered to be bioequivalent if the 90% confidence interval of AUC(0-infinity) for difference between both treatments fall in the range of 0.80-1.25; Ratio of Geometrical Mean = 1.059, 90% CI 2-sided [1.006 to 1.115]

2. Primary Outcome: AUC(0-infinity) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Statistical analysis of PK parameters was done using mixed effect model for evaluation of BE. Point estimate and associated adjusted 90% CI of difference between both the treatments were provided for AUC(0-infinity).
Time Frame: as for outcome 1
Population: BE analysis Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (90% Confidence Interval); unit: Hour*nanogram per milliliter
Groups:
- Paroxetine 40 mg, GSKT- Fasted: Eligible participants received a single dose of treatment A: GSKT, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in either treatment period 1 or 2 as per randomization under fasting condition.
- Paroxetine 40 mg, Mississauga- Fasted: Eligible participants received a single dose of treatment B: Mississauga, Paroxetine IR 40 mg (20 mg*2 tablets) administered orally on Day 1 in either treatment period 1 or 2 as per randomization under fasting condition.
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 36 | 36
Hour*nanogram per milliliter | 742.07 [615.82 to 894.21] | 745.22 [618.43 to 898.00]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fasted vs Paroxetine 40 mg, Mississauga- Fasted; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of Geometrical Mean = 0.996, 90% CI 2-sided [0.947 to 1.047]

3. Primary Outcome: Area Under the Concentration-time Curve From Administration Extrapolated to the Last Time of Quantifiable Concentration (AUC[0-t]) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Statistical analysis of PK parameters was done using mixed effect model for evaluation of BE. Point estimate and associated adjusted 90% CI of difference between both the treatments were provided for AUC(0-t).
Time Frame: as for outcome 1
Population: BE analysis Population
Measure: Geometric Mean (90% Confidence Interval); unit: Hour*nanogram per milliliter
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 41 | 41
Hour*nanogram per milliliter | 866.85 [733.56 to 1024.36] | 814.75 [689.47 to 962.80]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fed vs Paroxetine 40 mg, Mississauga- Fed; Test type: Equivalence — The two formulations were considered to be bioequivalent if the 90% confidence interval of AUC(0-t) for difference between both treatments fall in the range of 0.80-1.25; Ratio of Geometrical Mean = 1.064, 90% CI 2-sided [1.010 to 1.120]

4. Primary Outcome: AUC(0-t) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: as for outcome 3
Time Frame: as for outcome 1
Population: BE analysis Population
Measure: Geometric Mean (90% Confidence Interval); unit: Hour*nanogram per milliliter
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 37 | 37
Hour*nanogram per milliliter | 750.49 [623.30 to 903.64] | 753.83 [626.08 to 907.66]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fasted vs Paroxetine 40 mg, Mississauga- Fasted; Test type: Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of Geometrical Mean = 0.996, 90% CI 2-sided [0.949 to 1.044]

5. Primary Outcome: Maximum Observed Concentration (Cmax) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Statistical analysis of PK parameters was done using mixed effect model for evaluation of BE. Point estimate and associated adjusted 90% CI of difference between both the treatments were provided for Cmax.
Time Frame: as for outcome 1
Population: BE analysis Population
Measure: Geometric Mean (90% Confidence Interval); unit: Nanogram per milliliter
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 41 | 41
Nanogram per milliliter | 39.95 [35.36 to 45.14] | 39.02 [34.54 to 44.09]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fed vs Paroxetine 40 mg, Mississauga- Fed; Test type: Equivalence — The two formulations were considered to be bioequivalent if the 90% confidence interval of Cmax for difference between both treatments fall in the range of 0.80-1.25; Ratio of Geometrical Mean = 1.024, 90% CI 2-sided [0.952 to 1.101]

6. Primary Outcome: Cmax of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: as for outcome 5
Time Frame: as for outcome 1
Population: BE analysis Population.
Measure: Geometric Mean (90% Confidence Interval); unit: Nanogram per milliliter
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 37 | 37
Nanogram per milliliter | 36.86 [32.73 to 41.52] | 36.15 [32.10 to 40.72]
Statistical Analysis 1: Comparison: Paroxetine 40 mg, GSKT- Fasted vs Paroxetine 40 mg, Mississauga- Fasted; Test type: Equivalence — [test comment as in outcome 5, analysis 1]; Ratio of Geometrical Mean = 1.020, 90% CI 2-sided [0.968 to 1.074]

7. Secondary Outcome: Time to Reach Maximum Observed Concentration (Tmax) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Median and full range of Tmax have been presented.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. PK Population comprised of all randomized participants received at least one dose of study treatment and provided at least one evaluable PK concentration data. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 43 | 45
Hours | 5.00 [2.0 to 8.1] | 5.00 [2.0 to 8.0]

8. Secondary Outcome: Tmax of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: as for outcome 7
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (Full Range); unit: Hours
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 38 | 37
Hours | 5.00 [2.0 to 8.0] | 5.00 [2.0 to 8.1]

9. Secondary Outcome: Terminal Elimination Rate Constant (Lambda z) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Geometric mean and 95% CI of Lambda z have been presented.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 43 | 45
Per hour | 0.0433 [0.0385 to 0.0487] | 0.0462 [0.0422 to 0.0507]

10. Secondary Outcome: Lambda z of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: as for outcome 9
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Per hour
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 38 | 37
Per hour | 0.0483 [0.0444 to 0.0525] | 0.0494 [0.0451 to 0.0541]

11. Secondary Outcome: Terminal Elimination Half-life (t1/2) of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fed Condition
Description: Blood samples were collected at designated timepoints. PK parameters of Paroxetine were calculated using non-compartmental methods. Geometric mean and 95% CI have been presented.
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 43 | 45
Hours | 16.0002 [14.2232 to 17.9992] | 14.9913 [13.6850 to 16.4223]

12. Secondary Outcome: t1/2 of Paroxetine Following Single Oral Dose in Healthy Chinese Participants Under Fasting Condition
Description: as for outcome 11
Time Frame: as for outcome 1
Population: Pharmacokinetic Population. Only those participants with data available at the specified data points were analyzed.
Measure: Geometric Mean (95% Confidence Interval); unit: Hours
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 38 | 37
Hours | 14.3515 [13.2046 to 15.5980] | 14.0311 [12.8060 to 15.3734]

13. Secondary Outcome: Number of Participants With Non-serious Adverse Events and Serious Adverse Events (SAEs) Under Fed Condition
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement or events associated with liver injury and impaired liver function. Data has been presented treatment-wise.
Time Frame: Up to Day 26
Population: Safety Population. Safety Population comprised of all randomized participants who received at least one dose of study treatment. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 44 | 46
Participants
  Any non-SAEs | 14 | 13
  Any SAEs | 0 | 0

14. Secondary Outcome: Number of Participants With Non-SAE and SAEs Under Fasting Condition
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life-threatening, requires inpatient hospitalization or prolongation of existing hospitalization, results in persistent disability/incapacity, is a congenital anomaly/birth defect and other situations according to medical or scientific judgement or events associated with liver injury and impaired liver function. Data has been presented treatment-wise.
Time Frame: Up to Day 26
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 38 | 38
Participants
  Any non-SAEs | 12 | 16
  Any SAEs | 0 | 0

15. Secondary Outcome: Number of Participants With Chemistry Laboratory Values Relative to Potential Clinical Importance (PCI) Criteria on Day 16 Under Fed Condition
Description: Blood samples were collected to analyze the clinical chemistry laboratory parameters; alanine aminotransferase (ALT), albumin, alkaline phosphatase (ALP), aspartate aminotransferase (AST),calcium,creatinine, glucose, potassium (Pot) and sodium. PCI ranges were ALT (high: >=2 times upper limit of normal [ULN] units per liter [U/L]),albumin (low: <30 grams per liter),ALP (low: <20 international units per liter [IU/L] and high: >200 IU/L), AST (high: >=2 times ULN U/L),calcium (low: <2 millimoles per liter [mmol/L] and high: >2.75 mmol/L),creatinine (high: >133 micromoles per liter), glucose (low: <3 mmol/L and high: >9 mmol/L), Pot (low: <3 mmol/L and high: >5.5 mmol/L) and sodium (low: <130 mmol/L and high: >150 mmol/L). Participants were counted in the category that their value changed to (low, normal or high). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Data has been presented treatment-wise.
Time Frame: Day 16
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 22 | 22
Participants
  ALT, To low | 0 | 0
  ALT, To normal or no change | 22 | 22
  ALT, To high | 0 | 0
  Albumin, To low | 0 | 0
  Albumin, To normal or no change | 22 | 22
  Albumin, To high | 0 | 0
  ALP, To low | 0 | 0
  ALP, To normal or no change | 22 | 22
  ALP, To high | 0 | 0
  AST, To low | 0 | 0
  AST, To normal or no change | 22 | 22
  AST, To high | 0 | 0
  Calcium, To low | 0 | 0
  Calcium, To normal or no change | 22 | 22
  Calcium, To high | 0 | 0
  Creatinine, To low | 0 | 0
  Creatinine, To normal or no change | 22 | 22
  Creatinine, To high | 0 | 0
  Glucose, To low | 0 | 0
  Glucose, To normal or no change | 22 | 22
  Glucose, To high | 0 | 0
  Pot, To low | 0 | 0
  Pot, To normal or no change | 22 | 22
  Pot, To high | 0 | 0
  Sodium, To low | 0 | 0
  Sodium, To normal or no change | 22 | 22
  Sodium, To high | 0 | 0

16. Secondary Outcome: Number of Participants With Chemistry Laboratory Values Relative to PCI Criteria on Day 16 Under Fasting Condition
Description: Blood samples were collected to analyze the clinical chemistry laboratory parameters; ALT, albumin, ALP, AST, calcium, creatinine, glucose, Pot and sodium. PCI ranges were ALT (high: >=2 times ULN U/L), albumin (low: <30 grams per liter), ALP (low: <20 IU/L and high: >200 IU/L), AST (high: >=2 times ULN U/L), calcium (low: <2 mmol/L and high: >2.75 mmol/L), creatinine (high: >133 micromoles per liter), glucose (low: <3 mmol/L and high: >9 mmol/L), Pot (low: <3 mmol/L and high: >5.5 mmol/L) and sodium (low: <130 mmol/L and high: >150 mmol/L). Participants were counted in the category that their value changed to (low, normal or high). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Data has been presented treatment-wise.
Time Frame: Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Participants
  ALT, To low | 0 | 0
  ALT, To normal or no change | 19 | 19
  ALT, To high | 0 | 0
  Albumin, To low | 0 | 0
  Albumin, To normal or no change | 19 | 19
  Albumin, To high | 0 | 0
  ALP, To low | 0 | 0
  ALP, To normal or no change | 19 | 19
  ALP, To high | 0 | 0
  AST, To low | 0 | 0
  AST, To normal or no change | 19 | 19
  AST, To high | 0 | 0
  Calcium, To low | 0 | 0
  Calcium, To normal or no change | 19 | 19
  Calcium, To high | 0 | 0
  Creatinine, To low | 0 | 0
  Creatinine, To normal or no change | 19 | 19
  Creatinine, To high | 0 | 0
  Glucose, To low | 0 | 0
  Glucose, To normal or no change | 19 | 19
  Glucose, To high | 0 | 0
  Pot, To low | 0 | 0
  Pot, To normal or no change | 19 | 19
  Pot, To high | 0 | 0
  Sodium, To low | 0 | 0
  Sodium, To normal or no change | 19 | 19
  Sodium, To high | 0 | 0

17. Secondary Outcome: Number of Participants With Hematology Laboratory Values Relative to PCI Criteria on Day 16 Under Fed Condition
Description: Blood samples were collected to analyze; hematocrit(Hct),hemoglobin(Hb),erythrocytes and platelets. PCI ranges; Hct(Male[low: <0.03 proportion of red blood cells in blood and high: >0.54 proportion of red blood cells in blood] and Female[low: <0.04 proportion of red blood cells in blood and high: >0.54 proportion of red blood cells in blood]),Hb(Male [low: <110 grams per liter and high: >180 grams per liter) and Female[low: <100 grams per liter and high: >170 grams per liter]),erythrocytes(Male [low: <4.5x10^12 cells per liter and high: >5.5x10^12 cells per liter] and Female[low: <4 x10^12 cells per liter and high: >5 x10^12 cells per liter]) and platelets(low: <80x10^9 cells per liter and high: >400x10^9 cells per liter). Participants were counted in the category that their value changed to(low, normal or high). If values were unchanged(example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category.Data has been presented treatment-wise.
Time Frame: Day 16
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 22 | 22
Participants
  Erythrocytes, To low | 2 | 2
  Erythrocytes, To normal or no change | 20 | 19
  Erythrocytes, To high | 0 | 1
  Hct, To low | 0 | 0
  Hct, To normal or no change | 22 | 22
  Hct, To high | 0 | 0
  Hb, To low | 0 | 0
  Hb, To normal or no change | 22 | 22
  Hb, To high | 0 | 0
  Platelets, To low | 0 | 0
  Platelets, To normal or no change | 22 | 22
  Platelets, To high | 0 | 0

18. Secondary Outcome: Number of Participants With Hematology Laboratory Values Relative to PCI Criteria on Day 16 Under Fasting Condition
Description: Blood samples were collected to analyze; Hct, Hb, erythrocytes and platelets. PCI ranges were Hct (Male [low: <0.03 proportion of red blood cells in blood and high: >0.54 proportion of red blood cells in blood] and Female [low: <0.04 proportion of red blood cells in blood and high: >0.54 proportion of red blood cells in blood]), Hb (Male [low: <110 grams per liter and high: >180 grams per liter) and Female [low: <100 grams per liter and high: >170 grams per liter]), erythrocytes (Male [low: <4.5x10^12 cells per liter and high: >5.5x10^12 cells per liter] and Female [low: <4 x10^12 cells per liter and high: >5 x10^12 cells per liter]) and platelets (low: <80x10^9 cells per liter and high: >400x10^9 cells per liter). Participants were counted in the category that their value changed to (low, normal or high). If values were unchanged (example: High to High), or whose value became normal, were recorded in the 'To Normal or No Change' category. Data has been presented treatment-wise.
Time Frame: Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Participants
  Erythrocytes, To low | 1 | 0
  Erythrocytes, To normal or no change | 18 | 19
  Erythrocytes, To high | 0 | 0
  Hct, To low | 0 | 0
  Hct, To normal or no change | 19 | 19
  Hct, To high | 0 | 0
  Hb, To low | 0 | 0
  Hb, To normal or no change | 19 | 19
  Hb, To high | 0 | 0
  Platelets, To low | 0 | 0
  Platelets, To normal or no change | 19 | 19
  Platelets, To high | 0 | 0

19. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Method Under Fed Condition
Description: Urine samples were collected to assess urine occult blood, urine glucose, urine ketones, urine protein and monitor urine potential of hydrogen (pH). The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters (except urine pH) were recorded as negative and positive, indicating proportional concentrations in the urine sample. pH is a measure of hydrogen ion concentration and is used to determine the acidity or alkalinity of urine. Urine pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0). Dipstick test results for pH were presented as number of participants having pH value as 5, 6, 6.5, 7 or 8. Data has been presented treatment-wise.
Time Frame: Baseline (Day-7 to Day -1) and Day 16
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n=X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 22 | 25
Participants
  Glucose, Baseline, Negative, n=22,25 | 22 | 25
  Glucose, Baseline, Positive, n=22,25 | 0 | 0
  Glucose, Day 16, Negative, n=22,22: number analyzed (Participants) | 22 | 22
  Glucose, Day 16, Negative, n=22,22 | 22 | 22
  Glucose, Day 16, Positive, n=22,22: number analyzed (Participants) | 22 | 22
  Glucose, Day 16, Positive, n=22,22 | 0 | 0
  Ketones, Baseline, Positive, n=22,25 | 2 | 1
  Ketones, Baseline, Negative, n=22,25 | 20 | 24
  Ketones, Day 16, Positive,n=22,22: number analyzed (Participants) | 22 | 22
  Ketones, Day 16, Positive,n=22,22 | 1 | 0
  Ketones, Day 16, Negative,n=22,22: number analyzed (Participants) | 22 | 22
  Ketones, Day 16, Negative,n=22,22 | 21 | 22
  Occult blood, Baseline, Positive,n=22,25 | 2 | 3
  Occult blood, Baseline, Negative,n=22,25 | 20 | 22
  Occult blood, Day 16, Positive,n=22,22: number analyzed (Participants) | 22 | 22
  Occult blood, Day 16, Positive,n=22,22 | 5 | 3
  Occult blood, Day 16, Negative,n=22,22: number analyzed (Participants) | 22 | 22
  Occult blood, Day 16, Negative,n=22,22 | 17 | 19
  Protein, Baseline, Negative,n=22,25 | 22 | 25
  Protein, Baseline, Positive,n=22,25 | 0 | 0
  Protein, Day 16, Positive,n=22,22: number analyzed (Participants) | 22 | 22
  Protein, Day 16, Positive,n=22,22 | 1 | 0
  Protein, Day 16, Negative,n=22,22: number analyzed (Participants) | 22 | 22
  Protein, Day 16, Negative,n=22,22 | 21 | 22
  pH=5, Baseline,n=22,25 | 1 | 4
  pH=6, Baseline,n=22,25 | 7 | 5
  pH=6.5, Baseline,n=22,25 | 3 | 6
  pH=7, Baseline,n=22,25 | 9 | 10
  pH=8, Baseline,n=22,25 | 2 | 0
  pH=5, Day 16,n=22,22: number analyzed (Participants) | 22 | 22
  pH=5, Day 16,n=22,22 | 2 | 4
  pH=6, Day 16,n=22,22: number analyzed (Participants) | 22 | 22
  pH=6, Day 16,n=22,22 | 12 | 10
  pH=6.5, Day 16,n=22,22: number analyzed (Participants) | 22 | 22
  pH=6.5, Day 16,n=22,22 | 4 | 2
  pH=7, Day 16,n=22,22: number analyzed (Participants) | 22 | 22
  pH=7, Day 16,n=22,22 | 4 | 6
  pH=8, Day 16,n=22,22: number analyzed (Participants) | 22 | 22
  pH=8, Day 16,n=22,22 | 0 | 0

20. Secondary Outcome: Number of Participants With Urinalysis Results by Dipstick Method Under Fasting Condition
Description: Urine samples were collected to assess urine occult blood, urine glucose, urine ketones, urine protein and monitor urine pH. The dipstick test gave results in a semi-quantitative manner, and results for urinalysis parameters (except urine pH) were recorded as negative and positive, indicating proportional concentrations in the urine sample. pH is a measure of hydrogen ion concentration and is used to determine the acidity or alkalinity of urine. Urine pH is calculated on a scale of 0 to 14, values on the scale refer to the degree of alkalinity or acidity. A pH of 7 is neutral. A pH of less than 7 is acidic and a pH of greater than 7 is basic. Normal urine has a slightly acidic pH (5.0-6.0). Dipstick test results for pH were presented as number of participants having pH value as 5, 6, 6.5, 7 or 8. Data has been presented treatment-wise.
Time Frame: Baseline (Day-7 to Day -1) and Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Participants
  Glucose, Baseline, Negative, | 19 | 19
  Glucose, Baseline, Positive, | 0 | 0
  Glucose, Day 16, Negative, | 19 | 19
  Glucose, Day 16, Positive, | 0 | 0
  Ketones, Baseline, Negative | 19 | 19
  Ketones, Baseline, Positive | 0 | 0
  Ketones, Day 16,Positive | 1 | 1
  Ketones, Day 16, Negative | 18 | 18
  Occult blood, Baseline, Positive | 0 | 1
  Occult blood, Baseline, Negative | 19 | 18
  Occult blood, Day 16, Positive | 3 | 1
  Occult blood, Day 16, Negative | 16 | 18
  Protein, Baseline, Negative | 19 | 19
  Protein, Baseline, Positive | 0 | 0
  Protein, Day 16, Positive | 0 | 1
  Protein, Day 16, Negative | 19 | 18
  pH=5, Baseline | 3 | 2
  pH=6, Baseline | 2 | 3
  pH=6.5, Baseline | 5 | 4
  pH=7, Baseline | 6 | 9
  pH=8, Baseline | 3 | 1
  pH=5, Day 16 | 4 | 6
  pH=6, Day 16 | 13 | 11
  pH=6.5, Day 16 | 0 | 0
  pH=7, Day 16 | 2 | 2
  pH=8, Day 16 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for Electrocardiogram (ECG) Parameters Under Fed Condition
Description: A single 12-lead ECGs was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QT corrected (QTc) intervals. Clinically significant abnormal ranges were: heart rate: lower:<50 beats per minute and upper: >110 beats per minute; QT: Upper: >400 milliseconds (msec); QTc: Upper: >450 msec; PR: lower: <110 msec and upper: >220 msec; QRS: lower: <60 msec and upper: >120 msec. The number of participants with abnormal findings for ECG parameters have been presented. Data has been presented treatment-wise.
Time Frame: Baseline (Day-7 to Day -1) and Day 16
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 22 | 25
Participants
  Baseline, n=22, 25 | 0 | 0
  Day 16, n=22, 22: number analyzed (Participants) | 22 | 22
  Day 16, n=22, 22 | 1 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Abnormal Findings for ECG Parameters Under Fasting Condition
Description: A single 12-lead ECGs was obtained using an ECG machine that automatically calculates the heart rate and measures PR, QRS, QT and QTc intervals. Clinically significant abnormal ranges were: heart rate: lower :<50 beats per minute and upper: >110 beats per minute; QT: Upper: >400 msec; QTc: Upper: >450 msec; PR: lower: <110 msec and upper: >220 msec; QRS: lower: <60 msec and upper: >120 msec. The number of participants with abnormal findings for ECG parameters have been presented. Data has been presented treatment-wise.
Time Frame: Baseline (Day-7 to Day -1) and Day 16
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Participants
  Baseline | 0 | 0
  Day 16 | 0 | 0

23. Secondary Outcome: Diastolic Blood Pressure (DBP) and Systolic Blood Pressure (SBP) at Indicated Time-points Under Fed Condition
Description: Vital signs including DBP and SBP were measured at the indicated time-points and summarized during the study to evaluate the safety of the participants. Data has been presented treatment-wise.
Time Frame: Day 1 (post-dose), Day 2 (post-dose), Day 3, Day 4, Day 5, Day 11, Day 12 (pre-dose), Day 12 (post-dose), Day 13 (post-dose), Day 14, Day 15, Day 16
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 23 | 24
Millimeters of mercury
  DBP, Day 1 (post-dose), n=23,24 | 70.4 (9.27) | 67.8 (6.84)
  DBP, Day 2 (post-dose), n=23,24 | 69.0 (7.93) | 66.8 (7.38)
  DBP, Day 3, n=23,24 | 67.7 (7.11) | 64.5 (5.27)
  DBP, Day 4, n=23,24 | 67.5 (6.68) | 66.1 (6.86)
  DBP, Day 5, n=23,24 | 69.7 (6.98) | 68.9 (7.31)
  DBP, Day 11, n=21,22: number analyzed (Participants) | 21 | 22
  DBP, Day 11, n=21,22 | 69.9 (7.62) | 70.5 (8.98)
  DBP, Day 12 (pre-dose), n=21,22: number analyzed (Participants) | 21 | 22
  DBP, Day 12 (pre-dose), n=21,22 | 71.2 (6.59) | 72.7 (7.79)
  DBP, Day 12 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  DBP, Day 12 (post-dose), n=20,22 | 69.9 (7.71) | 72.2 (7.67)
  DBP, Day 13 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  DBP, Day 13 (post-dose), n=20,22 | 70.3 (6.50) | 72.9 (7.75)
  DBP, Day 14, n=20,22: number analyzed (Participants) | 20 | 22
  DBP, Day 14, n=20,22 | 70.3 (8.15) | 71.7 (7.09)
  DBP, Day 15, n=20,22: number analyzed (Participants) | 20 | 22
  DBP, Day 15, n=20,22 | 68.8 (6.14) | 70.4 (7.10)
  DBP, Day 16, n=20,22: number analyzed (Participants) | 20 | 22
  DBP, Day 16, n=20,22 | 72.8 (8.42) | 73.9 (6.65)
  SBP, Day 1 (post-dose), n=23,24 | 112.4 (10.13) | 111.8 (11.15)
  SBP, Day 2 (post-dose), n=23,24 | 113.8 (9.07) | 111.0 (10.19)
  SBP, Day 3, n=23,24 | 112.9 (9.46) | 109.4 (10.52)
  SBP, Day 4, n=23,24 | 111.1 (10.83) | 110.9 (10.97)
  SBP, Day 5, n=23,24 | 109.2 (10.31) | 109.8 (10.08)
  SBP, Day 11, n=21,22: number analyzed (Participants) | 21 | 22
  SBP, Day 11, n=21,22 | 109.0 (10.89) | 110.6 (9.18)
  SBP, Day 12 (pre-dose), n=21,22: number analyzed (Participants) | 21 | 22
  SBP, Day 12 (pre-dose), n=21,22 | 107.2 (9.54) | 108.5 (8.34)
  SBP, Day 12 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  SBP, Day 12 (post-dose), n=20,22 | 112.4 (9.66) | 112.4 (11.42)
  SBP, Day 13 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  SBP, Day 13 (post-dose), n=20,22 | 111.4 (10.18) | 112.0 (8.80)
  SBP, Day 14, n=20,22: number analyzed (Participants) | 20 | 22
  SBP, Day 14, n=20,22 | 107.0 (9.49) | 105.5 (8.44)
  SBP, Day 15, n=20,22: number analyzed (Participants) | 20 | 22
  SBP, Day 15, n=20,22 | 107.3 (7.73) | 106.0 (9.62)
  SBP, Day 16, n=20,22: number analyzed (Participants) | 20 | 22
  SBP, Day 16, n=20,22 | 107.1 (8.94) | 105.9 (6.29)

24. Secondary Outcome: DBP and SBP at Indicated Time-points Under Fasting Condition
Description: as for outcome 23
Time Frame: as for outcome 23
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Millimeters of mercury
  DBP, Day 1 (post-dose) | 71.8 (6.37) | 70.9 (6.56)
  DBP, Day 2 (post-dose) | 68.3 (7.59) | 68.7 (7.61)
  DBP, Day 3 | 66.2 (6.99) | 67.8 (9.22)
  DBP, Day 4 | 68.3 (8.29) | 68.8 (5.91)
  DBP, Day 5 | 68.1 (6.16) | 73.3 (7.31)
  DBP, Day 11 | 71.9 (6.62) | 71.4 (7.36)
  DBP, Day 12 (pre-dose) | 72.6 (8.00) | 71.2 (9.11)
  DBP, Day 12 (post-dose) | 73.5 (6.29) | 70.3 (7.59)
  DBP, Day 13 (post-dose) | 72.6 (6.72) | 69.6 (7.22)
  DBP, Day 14 | 72.2 (6.96) | 70.2 (4.76)
  DBP, Day 15 | 70.6 (7.65) | 68.7 (8.39)
  DBP, Day 16 | 71.9 (7.32) | 71.1 (8.28)
  SBP, Day 1 (post-dose) | 107.4 (10.56) | 109.2 (10.82)
  SBP, Day 2 (post-dose) | 108.1 (11.85) | 110.1 (10.13)
  SBP, Day 3 | 106.3 (10.19) | 108.2 (12.21)
  SBP, Day 4 | 105.1 (10.31) | 107.4 (8.78)
  SBP, Day 5 | 104.4 (9.17) | 111.3 (12.03)
  SBP, Day 11 | 113.2 (13.72) | 111.4 (12.88)
  SBP, Day 12 (pre-dose) | 108.3 (10.40) | 107.4 (9.63)
  SBP, Day 12 (post-dose) | 111.6 (9.63) | 107.5 (8.84)
  SBP, Day 13 (post-dose) | 111.7 (10.50) | 109.9 (11.86)
  SBP, Day 14 | 110.5 (12.18) | 104.5 (9.48)
  SBP, Day 15 | 108.5 (10.56) | 107.4 (9.63)
  SBP, Day 16 | 110.7 (12.70) | 104.2 (9.65)

25. Secondary Outcome: Pulse Rate (PR) at Indicated Time-points Under Fed Condition
Description: Vital sign including PR was measured at the indicated time-points and summarized during the study to evaluate the safety of the participants. Data has been presented treatment-wise.
Time Frame: as for outcome 23
Population: as for outcome 19
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 23 | 24
Beats per minute
  Day 1 (post-dose), n=23,24 | 72.3 (10.57) | 72.0 (8.83)
  Day 2 (post-dose), n=23,24 | 72.8 (8.22) | 74.1 (9.98)
  Day 3, n=23,24 | 74.0 (9.11) | 75.8 (10.07)
  Day 4, n=23,24 | 75.5 (7.13) | 75.7 (11.02)
  Day 5, n=23,24 | 68.7 (7.03) | 68.3 (8.87)
  Day 11, n=21,22: number analyzed (Participants) | 21 | 22
  Day 11, n=21,22 | 75.0 (11.05) | 77.7 (8.38)
  Day 12 (pre-dose), n=21,22: number analyzed (Participants) | 21 | 22
  Day 12 (pre-dose), n=21,22 | 65.8 (9.00) | 64.7 (7.57)
  Day 12 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  Day 12 (post-dose), n=20,22 | 72.8 (10.85) | 76.2 (10.15)
  Day 13 (post-dose), n=20,22: number analyzed (Participants) | 20 | 22
  Day 13 (post-dose), n=20,22 | 73.7 (11.86) | 73.8 (8.07)
  Day 14, n=20,22: number analyzed (Participants) | 20 | 22
  Day 14, n=20,22 | 75.6 (10.72) | 77.6 (9.88)
  Day 15, n=20,22: number analyzed (Participants) | 20 | 22
  Day 15, n=20,22 | 77.5 (11.33) | 75.5 (8.38)
  Day 16, n=20,22: number analyzed (Participants) | 20 | 22
  Day 16, n=20,22 | 69.4 (8.54) | 72.6 (9.51)

26. Secondary Outcome: Pulse Rate (PR) at Indicated Time-points Under Fasting Condition
Description: as for outcome 25
Time Frame: as for outcome 23
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Beats per minute
  Day 1 (post-dose) | 65.4 (8.80) | 67.5 (7.19)
  Day 2 (post-dose) | 74.8 (7.40) | 75.3 (8.31)
  Day 3 | 74.9 (8.45) | 77.2 (10.69)
  Day 4 | 74.2 (8.74) | 72.8 (9.86)
  Day 5 | 67.3 (6.82) | 71.2 (9.60)
  Day 11 | 81.8 (9.72) | 84.1 (9.20)
  Day 12 (pre-dose) | 66.5 (8.73) | 66.8 (10.48)
  Day 12 (post-dose) | 67.5 (8.96) | 65.2 (7.19)
  Day 13 (post-dose) | 78.1 (11.03) | 75.4 (7.54)
  Day 14 | 78.9 (11.12) | 76.8 (8.25)
  Day 15 | 78.2 (8.38) | 75.9 (9.58)
  Day 16 | 75.7 (10.39) | 71.3 (7.92)

27. Secondary Outcome: Respiratory Rate (RR) at Indicated Time-point Under Fed Condition
Description: Vital sign including RR was measured at the indicated time-point and summarized during the study to evaluate the safety of the participants. Data has been presented treatment-wise.
Time Frame: Day 11
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 21 | 22
Breaths per minute | 17.8 (1.78) | 18.6 (1.79)

28. Secondary Outcome: RR at Indicated Time-point Under Fasting Condition
Description: as for outcome 27
Time Frame: Day 11
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Breaths per minute | 19.2 (1.38) | 19.4 (1.16)

29. Secondary Outcome: Temperature at Indicated Time-point Under Fed Condition
Description: Vital sign including temperature was measured at the indicated time-point and summarized during the study to evaluate the safety of the participants. Data has been presented treatment-wise.
Time Frame: Day 11
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed
Number analyzed (Participants) | 21 | 22
Celsius | 36.70 (0.307) | 36.59 (0.333)

30. Secondary Outcome: Temperature at Indicated Time-point Under Fasting Condition
Description: as for outcome 29
Time Frame: Day 11
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Celsius
Arm/Group | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
Number analyzed (Participants) | 19 | 19
Celsius | 36.84 (0.187) | 36.74 (0.256)

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and non-serious AEs were collected from the start of study treatment up to Day 26.
Description: SAEs and Non-SAEs were reported as per the treatment for the Safety Population which comprised of all randomized participants who received at least 1 dose of study treatment.
Arm/Group | Paroxetine 40 mg, GSKT- Fed | Paroxetine 40 mg, Mississauga- Fed | Paroxetine 40 mg, GSKT- Fasted | Paroxetine 40 mg, Mississauga- Fasted
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/46 | 0/38 | 0/38
Serious Adverse Events (participants affected / at risk) | 0/44 | 0/46 | 0/38 | 0/38
Other Adverse Events (participants affected / at risk) | 14/44 | 13/46 | 12/38 | 16/38
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Paroxetine 40 mg, GSKT- Fed (N=44) | Paroxetine 40 mg, Mississauga- Fed (N=46) | Paroxetine 40 mg, GSKT- Fasted (N=38) | Paroxetine 40 mg, Mississauga- Fasted (N=38)
Bacterial test (Investigations) | 1 | 1 | 2 | 1
White blood cells urine positive (Investigations) | 1 | 1 | 3 | 3
Alanine aminotransferase increased (Investigations) | 1 | 0 | 0 | 0
Blood uric acid increased (Investigations) | 1 | 0 | 0 | 0
Blood urine present (Investigations) | 1 | 0 | 0 | 0
Occult blood positive (Investigations) | 1 | 0 | 0 | 0
White blood cell count decreased (Investigations) | 0 | 3 | 1 | 0
Bilirubin conjugated increased (Investigations) | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 1 | 1 | 0
Blood glucose decreased (Investigations) | 0 | 1 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 2 | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 1 | 5 | 6
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 2
Toothache (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Mouth swelling (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 0 | 0 | 5
Dizziness (Nervous system disorders) | 1 | 0 | 6 | 4
Rash (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0
Cold sweat (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 0
Vision blurred (Eye disorders) | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 0 | 1 | 0
Mean cell haemoglobin decreased (Investigations) | 0 | 0 | 1 | 0
Mean cell volume decreased (Investigations) | 0 | 0 | 1 | 0
White blood cell count increased (Investigations) | 0 | 0 | 1 | 0
Bacterial test positive (Investigations) | 0 | 0 | 0 | 2
Protein urine present (Investigations) | 0 | 0 | 0 | 1
Urine ketone body present (Investigations) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Statistical Analysis Plan (2018-09-06): https://cdn.clinicaltrials.gov/large-docs/73/NCT03329573/SAP_001.pdf
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT03329573/Prot_002.pdf